CLINICAL TRIAL: NCT05720767
Title: A Phase 1, Open-label, 2-Part, 2-Period Fixed-Sequence Crossover Study to Assess the Effect of Itraconazole, and the Effect of Rifampin on the Pharmacokinetics of HMPL-523 in Healthy Volunteers
Brief Title: HMPL-523 CYP3A/P-gp Inhibitor and CYP Inducer Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-523-00US2
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Relapsed or Refractory Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma | interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A - Itraconazole (Experimental): HMPL-523 will be supplied as 100 and 150 mg tablets and will be administered PO as a single dose of 400 mg (combination of 2 of 150 mg tablets and 1 of 100 mg tablet) on two separate occasions (Day 1 and Day 10) in Part A. Itraconazole will be supplied as 100 mg capsules and will be administered as doses of 200 mg (2 × 100 mg) PO BID on Day 6 and 200 mg PO QD on Days 7 to 14 in Part A.
  Interventions: Drug: HMPL-523; Drug: Itraconazole
- Part B - Rifampin (Experimental): HMPL-523 will be supplied as 100 and 150 mg tablets and will be administered PO as a single dose of 700 mg (combination of 4 of 150 mg tablets and 1 of 100 mg tablet) on two separate occasions (Day 1 and Day 13) in Part B. Rifampin will be supplied as 300 mg capsules and will be administered as doses of 600 mg (2 × 300 mg) PO QD on Days 6 to 17 in Part B.
  Interventions: Drug: HMPL-523; Drug: Rifampin

INTERVENTIONS:
Drug: HMPL-523 — HMPL-523 is a selective small-molecule SYK inhibitor.
Drug: Itraconazole — Itraconazole is an FDA approved synthetic triazole antifungal agent
  Arms: Part A - Itraconazole
Drug: Rifampin — Rifampin is an FDA approved semisynthetic antiobiotic derivative indicated in the treatment of both tuberculosis and meningococcal carrier state
  Arms: Part B - Rifampin

SUMMARY:
A Phase 1, Open-label, 2-Part, 2-Period Fixed-Sequence Crossover Study to Assess the Effect of Itraconazole, a CYP3A and P-glycoprotein Inhibitor, and the Effect of Rifampin, a CYP Enzyme Inducer, on the Pharmacokinetics of HMPL-523 in Healthy Volunteers

DETAILED DESCRIPTION:
This study will be a single-center, open-label, 2-part, 2-period fixed-sequence crossover study to be conducted with 28 healthy male and female volunteers. The study will consist of a Screening Phase (Screening and Day -1), a Treatment Phase (Period 1 and Period 2), and an End of Study (EOS) Phase.

ELIGIBILITY:
Inclusion Criteria:

* 1. The volunteer is male or female between the ages of 18 and 55 years old (inclusive) at the time of informed consent.

  2. The volunteer has a body mass index (BMI) >18 and ≤29.9 kg/m2 at screening.

  3. Females must be postmenopausal (defined as absence of menses for at least one year without alternative medical cause) or permanently sterile by total hysterectomy, bilateral oophorectomy, or bilateral salpingectomy.

  4. Males, including those who have had a successful vasectomy, must use a condom during sexual intercourse with women of childbearing potential, starting from their first dose of study drug through 30 days after their last dose of study drug. Alternatively, abstinence is allowed if it is the normal and preferred lifestyle of the volunteer.

  5. The volunteer must provide written informed consent prior to any study specific screening procedures.

  6. The volunteer is willing and able to comply with all aspects of the protocol, as determined by the PI.

  7. The volunteer must have normal laboratory results for total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT); creatinine clearance must be > 90 mL/min estimated using the Cockcroft-Gault equation.

Exclusion Criteria:

* 1. The volunteer has a known history of any gastrointestinal surgery or any condition possibly affecting drug absorption (eg, cholecystectomy, gastrectomy, achlorhydria, peptic ulcer disease, or history of stomach or intestinal surgery or resection).

Note: Appendectomy and hernia repairs are allowed.

2. The volunteer had a clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to the first dose.

3. The volunteer has evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at screening or at Day -1 check-in (baseline).

4. The volunteer has systolic blood pressure >140 mmHg or a diastolic blood pressure >90 mmHg.

5. The volunteer has a clinically significant ECG abnormality, including a marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTcF interval >450 msec), or had a family history of prolonged QTc syndrome or sudden death.

6. The volunteer has a history of smoking or use of nicotine-containing substances within the previous 2 months, as determined by medical history or volunteer's verbal report and confirmed by cotinine test at check-in for each treatment period.

7. The volunteer has a history of drug or alcohol misuse within 6 months prior to screening or a positive urine drug test at screening or at check-in for each treatment period.

8. The volunteer has been diagnosed with acquired immune deficiency syndrome or has performed tests that are positive for human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).

9. The volunteer has participated in a clinical trial of another study drug before screening, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks, whichever is longer, or the volunteer is currently enrolled in another clinical trial.

10. The volunteer has consumed grapefruit, starfruit, Seville oranges, or their products within 7 days prior to the first dose.

11. The volunteer has consumed herbal preparations/medications, including, but not limited to, St. John's Wort, kava, ephedra (ma huang), Ginkgo biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng, within 7 days prior to the first dose (21 days for St. John's Wort).

12. The volunteer has experienced a weight loss or gain of >10% within 4 weeks prior to the first dose as noted by medical history and weight at screening and check-in.

13. The volunteer has received blood or blood products within 4 weeks, donated blood or blood products within 8 weeks prior to the first dose or donated double red cell within 16 weeks prior to first dose.

14. The volunteer has used any over-the-counter (OTC) medications or prescription drugs (including medications that can lower gastric acid, inhibit or induce P-gp and/or CYP3A4) within 5 half-lives of these drugs or 2 weeks prior to the first dose of study drug, whichever is longer.

15. The volunteer is allergic to any of the study drugs (or its excipients) to be given in this study.

16. A female participant is pregnant, lactating, or breastfeeding.

17. A male volunteer who plans to donate sperm or father a child within 30 days after receiving the study drug.

18. The volunteer has any condition that would make him or her, in the opinion of the PI or Sponsor, unsuitable for the study, or who, in the opinion of the PI, is not likely to complete the study for any reason.

Note: One repeat of laboratory assessments may be performed at screening and at Check-In (Day -1) at the discretion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
PK parameter for HMPL-523: AUC0-t | Day 1 to 18
  Area under the plasma concentration-time curve from time 0 to time of the last measurable concentration
PK parameter for HMPL-523: AUC0-inf | Day 1 to 18
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity (if data permit)
PK parameter for HMPL-523: Cmax | Day 1 to 18
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Incidence of Adverse Events/ Serious Adverse Events | Day 1 to Day 18
  Any untoward medical occurrence associated with the study drug

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No